CLINICAL TRIAL: NCT03429361
Title: Testing the Value of Smartphone Assessments of People With Mood Disorders: A Pilot, Exploratory, Longitudinal Study
Brief Title: Testing the Value of Smartphone Assessments of People With Mood Disorders
Status: Completed | Type: Observational
Sponsor: Mindstrong (Industry)
Collaborators: Kadima Neuropsychiatry Institute (Other)
Responsible Party: Sponsor
Other Study IDs: 17-01
Record Dates: First submitted 2018-01-23; First posted 2018-02-12 (Actual); Last update posted 2019-08-22 (Actual); Status verified 2019-08

CONDITIONS: Major Depressive Disorder; Bipolar Disorder
MeSH Terms: conditions — Depressive Disorder, Major; Bipolar Disorder

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Health by Mindstrong — Health by Mindstrong is a smartphone application that collects data on a participant's smartphone usage patterns.

SUMMARY:
The purpose of this study is two-fold:

1. To identify the best smartphone data features (based on keyboard, sensor, voice/speech data) that correlate with mood, anxiety, and cognitive assessments in patients with Major Depressive Disorder (MDD) and Bipolar Depression (BD).
2. To identify the best smartphone data features (based on keyboard, sensor, voice/speech at a) that predict relapse and remission in MDD or BD.

DETAILED DESCRIPTION:
Progress in psychiatry will require better measurement. Currently, few clinicians use standard rating instruments for either diagnosis or outcomes. As a result, clinicians often fail to detect when a patient is not improving and fail to adjust treatments accordingly. Yet even with the use of standard rating instruments, there are serious shortcomings because they are used episodically, usually in an office environment, and they rely solely on subjective reports. Given the importance of objective measures of mood, anxiety, and cognition, it is critical for clinicians and patients to have better assessments if we are to achieve better mental healthcare.

The advent of smartphones provides a potential solution for the lack of objective measurement. The wide use of phones gives us the opportunity to collect passive, objective, continuous data relevant to mood, anxiety, and cognition. While several studies have demonstrated the feasibility of digital phenotyping psychiatric patients, the clinical value of this approach has yet to be demonstrated.

Stated simply the question is: can the data from a smartphone be used in clinical practice to improve care? Specifically, will sensor data, keyboard behavior, or voice and speech metrics yield features that can be validated with clinical assessments? Can these features identify relapse and remission even before clinical change is apparent with traditional ratings? Will this information alter care and improve outcomes? This pilot investigation is designed to answer the questions about validation and prediction by studying mood changes in patients treated with ketamine, a rapid-acting antidepressant. The final question about care and outcomes will be addressed separately.

Thus, the current study is a 6 month open, exploratory study that follows longitudinally patients with MDD or BD who are receiving outpatient treatment at the Kadima Clinic. The Kadima Clinic is a private outpatient mental health service providing a range of treatments for people with mood disorders. All patients will be receiving ketamine treatment in the Kadima Clinic; however, this is a study of smartphone features as digital biomarkers, not a study of ketamine efficacy or safety. While the ketamine treatment will not be the focus of this study, its rapid efficacy yields an ideal opportunity for testing and tuning the Mindstrong digital phenotyping app. There will not be randomization, use of placebo, or administration of blinded medication. Patients will be selected based on their willingness to participate in clinical assessments and their use of a smartphone.

The design includes screening and assessment during the week prior to treatment and follow-up at regular intervals for at least 3 weeks and no more than 6 months following treatment. Assessments will be completed by the patient, by a trained clinical rater, and by a significant other.

After completing the enrollment consent, the Mindstrong application (app) is installed in each participant's smartphone. The app is resident on the participant's mobile phone for 6 months. The participant can at any time choose to uninstall the app. The Mindstrong app unobtrusively monitors the participant's use of the mobile phone. The data captured by the app is transmitted over secure channel to a secure data storage site on Amazon Web Services (AWS) cloud infrastructure. All data captured by the app is encrypted.

ELIGIBILITY:
Inclusion Criteria:

* Adult male or female aged 18 to 65 years (inclusive) at time of informed consent
* Diagnosis of Major Depression Disorder (MDD) or Bipolar Disorder (BD) as assessed using the Structured Clinical Interview for DSM Disorders-Clinical Trials (SCID-CT)
* Montgomery-Asberg Depression Rating Scale (MADRS) ≥ 26; Patient Health Questionnaire (PHQ-9) ≥ 15; Clinical Global Impression (CGI) ≥ 4 at screening
* Ownership of a personal smartphone and willingness to install and maintain the Mindstrong app for digital assessments throughout participation in the study
* Able to understand and comply with instructions in English
* Has a significant other who accompanies participant to treatment appointments and agrees to complete assessments
* Undergoing ketamine treatment at the Kadima Clinic, or determined by the Kadima Clinic to be eligible for ketamine treatment and agrees to receive such treatment prior to being asked to participate in this research

Exclusion Criteria:

* Female who is currently pregnant or planning a pregnancy within 6 months
* Has any other current Axis I DSM-5 disorder other than MDD or BD, which is the primary focus of treatment
* Has any other clinically significant medical condition or circumstance that, in the opinion of the Investigator, could affect patient safety, preclude evaluation of response, interfere with the ability to comply with study procedures, or prohibit completion of the study
* Has a visual or physical motor impairment that could interfere with study tasks
* Is site personnel directly affiliated with this study

Ages: 18 Years to 65 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: The study population includes men and women between the ages of 18 and 65 years, with a diagnosis of Major Depressive Disorder (MDD) or Bipolar Disorder (BD), currently undergoing ketamine treatment for that disorder.
Sampling Method: Non-Probability Sample
Enrollment: 23 (Actual)
Dates: Start 2017-08-08 (Actual); Primary Completion 2019-05-30 (Actual); Study Completion 2019-05-30 (Actual)

PRIMARY OUTCOMES:
Hamilton Depression Rating Scale (HAM-D) | 6 months
  A repeated measures, within-subject design using exploratory techniques will identify the best smartphone usage features or combination of features that correlate with or predict change on the HAM-D at post-treatment and follow-up.
Cognitive Battery | 6 months
  Cognitive Battery includes: Self-report emotional referent task, face-morph task, dot-probe task, choice reaction time, forward digit span, Trails A&B, digit-symbol substitution test, delayed memory recall, Stroop, Conners Continuous Performance Test, 2-Back test.
  A repeated measures, within-subject design using exploratory techniques will identify the best smartphone usage features or combination of features that correlate with or predict change on the Cognitive Battery at post-treatment and follow-up.
Hamilton Anxiety Rating Scale (HAM-A) | 6 months
  A repeated measures, within-subject design using exploratory techniques will identify the best smartphone usage features or combination of features that correlate with or predict change on the HAM-A at post-treatment and follow-up.
Patient Health Questionnaire (PHQ-9) | 6 months
  A repeated measures, within-subject design using exploratory techniques will identify the best smartphone usage features or combination of features that correlate with or predict relapse, defined as PHQ-9 > 20 and/or 67% reduction in PHQ-9 improvement between baseline and post-treatment or follow-up, at post-treatment and follow-up.

CONTACTS AND LOCATIONS:
Overall Officials: Paul Dagum, MD PhD, Principal Investigator — Mindstrong; David Feifel, MD PhD, Principal Investigator — Kadima Neuropsychiatry Institute
Locations (1):
- Kadima Neuropsychiatry Institute, La Jolla, California, United States

IPD SHARING:
Plan to Share IPD: Undecided